CLINICAL TRIAL: NCT04850014
Title: Physiologically-based Pharmacokinetic Modelling Applied to Acetaminophen- Poisoned Obese Children
Brief Title: PBPK Modelling Applied to Acetaminophen Poisoned Obese Children
Acronym: IntoxPara
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1244
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Poisoning; Obesity
Keywords: PBPK; Modelling; Acetaminophen; Paracetamol; Pediatrics; Obesity; Pharmacokinetics; Toxicokinetics; Poisoning
MeSH Terms: conditions — Poisoning; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Poisoned patients: All subjects with paracetamolemia in the context of paracetamol poisoning
  Interventions: Other: Anthropomorphism; Other: Relevant clinical datas
- Control group: Acetaminophen-poisoned patient being non-obese
  Interventions: Other: Anthropomorphism; Other: Relevant clinical datas

INTERVENTIONS:
Other: Anthropomorphism — Height, weight, body surface area, body mass index, exact age (date of birth or age in days, months and years), falling which year of birth gender
Other: Relevant clinical datas — Medical history Concomitant medication Paracetamol intake : dosage, delay, context, route of intake Alcohol intake Smoking status (including active and passive exposition or no exposition) Curative treatment / Antidote / purifying treatment received and time of introduction Clinical signs, Acetaminophen concentration in plasma with associated accurate time of sampling (date, hour and time following acetaminophen intake Liver and kindney function assessment by measure measuring plasma concentration of: AST, ALT, Factor V, Prothrombin, APTT, INR, albuminemia, bilirubin, phosphorus, pH, creatitine. And GFR estimation.
  Imaging.

SUMMARY:
Childhood obesity is increasing globally. Changes in body composition and physiology in obesity setting modify pharmacokinetic parameters and might increase the risk in case of poisoning. Acetaminophen is a drug often implied in poisoning in children population, especially in adolescent attempting suicide. In practice, clinicians use weight to assess intoxication severity, but depending on the weight chosen (actual weight, lean body weight, ideal weight,..) the severity assessment can change as well as medical care needed. In this context we hypothesize that a PBPK modelling would be helpful to predict toxic dosing in obese population and especially in obese adolescent or children. The primary objective of this study is to collect data related to acetaminophen-poisoned patient with at least one acetaminophen concentration sampling and whose clinical outcome is known in order to refine and validate such a PBPK model.

ELIGIBILITY:
Inclusion Criteria:

* All subjects >/= 10 year old
* Availability of at least one positive acetaminophen concentration with its associated sampling time
* Known clinical outcome

Exclusion Criteria:

* < 10 year old
* lack of data-

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Poisoned acetaminophen subjects
  * At least one acetaminophen blood sample result available in data base
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Acetaminophen concentration | 31 october 2021
  With hour post-ingestion provided

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France